CLINICAL TRIAL: NCT02832648
Title: The Effect of Selenium Supplementation on Musculoskeletal Health in Older Women Double-blind, Randomised, Placebo-controlled Trial
Brief Title: Selenium for Musculoskeletal Health
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STH19102; NIHR EME 14-200-20 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- selenase 200mcg (Experimental): selenium as selenase 200mcg once daily, oral
  Interventions: Dietary Supplement: selenase (selenium)
- selenase 50mcg (Experimental): selenium as selenase 50mcg once daily, oral
  Interventions: Dietary Supplement: selenase (selenium)
- placebo (Placebo Comparator): matched placebo, once daily, oral
  Interventions: Dietary Supplement: selenase (selenium)

INTERVENTIONS:
Dietary Supplement: selenase (selenium) — Selenase (Biosyn, Germany) Sodium selenite pentahydrate

SUMMARY:
This research aims to determine whether selenium supplements improve bone and muscle health in older women at risk of osteoporosis (low bone density or weak bones) and fracture (broken bones).

Osteoporosis is a major public health problem. One in two women and one in five men over age 50 will have a fracture. Fractures cause pain, disability and reduce life-expectancy. Women with below-average bone density around the time of the menopause might have previously taken hormone replacement (HRT) to prevent osteoporosis, but HRT is much less used now due to side effects. Therefore there is a need for safe, effective and inexpensive preventative interventions for women at risk of osteoporosis.

Selenium is a chemical nutrient present in several human proteins, including anti-oxidants. Anti-oxidants may protect against ageing of tissues, including bone, by mopping up damaging reactive oxygen molecules (sometimes called 'free radicals'). Selenium is present in soil, and so is obtained from many foods. However, soil selenium levels are low in Europe, and dietary intake in the UK is below recommended levels.

We previously found that women with higher blood selenium levels have stronger bones, but this doesn't prove that giving selenium will improve bone strength.

The investigators propose a randomised controlled trial to compare selenium supplements with a placebo (dummy treatment) in women with below-average bone density. The investigators will give selenium (at two different doses) or placebo to 120 women for six months and use blood and urine tests and bone density scans to see if giving selenium does have any effect on bone. The investigators will also do muscle function tests and measurements of free radical molecules.

DETAILED DESCRIPTION:
This is a double-blind, randomised, placebo controlled trial. We will evaluate two doses of selenium (50 and 200mcg) vs placebo over six months.

Participants are postmenopausal women with osteopenia or osteoporosis (T-score -1.0 to -3.0).

The investigators will include participants with any baseline serum selenium concentration for generalisability, but the primary endpoint efficacy analysis will only include women with baseline serum selenium below 120 mcg/l.

Primary endpoint: Urinary N-telopeptide of type I collagen (NTX/Cr). Secondary endpoints: other bone turnover markers, BMD, muscle function, thyroid function, blood glucose, anti-oxidant activity, inflammatory markers The investigators will make the primary analysis based on women with baseline serum selenium below 120 mcg/l. To ensure adequate power for this analysis we will plan to recruit 120 women (we expect that 100 of the 120 will have serum selenium below 120 mcg/l based on our previous cross-sectional study). The investigators will review the baseline serum selenium results when 40 women have been recruited to confirm the expected distribution of baseline levels, and we will adjust the total recruitment number accordingly to ensure at least 99 women with serum selenium below 120mcg/l have been randomised for the final primary endpoint intention-to-treat analysis.

Participants will be randomised according to a schedule produced by Sheffield Teaching Hospitals pharmacy according to their standard operating procedure. Randomisation will be carried out independently of the study investigators using block randomisation. The blind will only be broken if judged by the PI as clinically necessary for the wellbeing of a participant.

The study may be stopped early if the investigators, sponsor or DMEC identify a safety concern.

Trial management will be done by the Academic Unit of Bone Metabolism CTIMP group (who meet monthly), and progress reported to the AUBM management group and Lay Panel. We will establish a TSC and DMEC.

ELIGIBILITY:
Inclusion Criteria:

women age over 55y at least 5y postemenopausal willing and able to give informed consent lumbar spine or total hip BMD T-score between -1.0 and -3.0 not clinically requiring treatment for osteoporosis

Exclusion Criteria:

diabetes mellitus, thyroid dysfunction, any conditions known to affect bone metabolism (such as inflammatory disease, parathyroid disease, malabsorption ), medications known to affect bone metabolism (such as osteoporosis treatment, aromatase inhibitors, anti-epileptics), alcohol intake >21 units per week, prolonged immobility (>3 months), fracture in the last year, taken selenium supplements in the last year

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
urine NTX (N-terminal cross-linking telopeptide of type I collagen) | 6 months
  bone resorption marker

SECONDARY OUTCOMES:
serum selenium and selenoprotein P | 6 months
  measures of selnium status
other biochemical markers of bone turnover | 6 months
  CTX (C-terminal cross-linking telopeptide of type I collagen), osteocalcin, PINP (Procollagen type I N propeptide)
bone mineral density | 6m
  DXA lumbar spine and total hip
physical function | 6m
  short physical performance battery and hand grip strength
anti-oxidant activity | 6m
  glutathione peroxidase, hydroperoxide, reactive oxygen species
inflammatory markers | 6m
  serum interleukin-6, highly senetive c-reative protein
serum insulin and glucose ratio | 3m, 6m
  safety monitoring for diabetes
thyroid stimulating hormone | 3m, 6m
  safety monitoring for thyroid dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Walsh, MbChB PhD, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walsh JS, Jacques RM, Schomburg L, Hill TR, Mathers JC, Williams GR, Eastell R. Effect of selenium supplementation on musculoskeletal health in older women: a randomised, double-blind, placebo-controlled trial. Lancet Healthy Longev. 2021 Apr;2(4):e212-e221. doi: 10.1016/S2666-7568(21)00051-9. PMID 33842907

DOCUMENTS (1):
  • Study Protocol (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT02832648/Prot_000.pdf